CLINICAL TRIAL: NCT01364194
Title: Periarticular Injection With Bupivacaine For Post-Operative Pain Control In Total Knee Replacement: A Prospective Randomized Double-Blind Controlled Trial
Brief Title: Local Infiltration With Bupivacaine to Increase Quality of Post-operative Pain Control in Total Knee Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Keerati Chareancholvanich, MD, Siriraj Hospital, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 516/2552(EC3)
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Pain, Postoperative; Arthropathy of Knee Joint
Keywords: Post operative pain; Total knee replacement; Total knee arthroplasty; Bupivacaine; Periarticular injection; Placebo; Morphine consumption
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.25% Bupivacaine (Active Comparator): Periarticular injection with 20 ml of 0.25% bupivacaine before wound closure.
  Interventions: Drug: 0.25% Bupivacaine
- 0.9% normal saline (Placebo Comparator): Periarticular injection with 20 ml of 0.9% normal saline before wound closure.
  Interventions: Drug: 0.9% normal saline

INTERVENTIONS:
Drug: 0.25% Bupivacaine — Periarticular injection with 20 ml of 0.25% bupivacaine before wound closure.
  Other Names: Marcaine
  Arms: 0.25% Bupivacaine
Drug: 0.9% normal saline — Periarticular injection with 20 ml of 0.9% normal saline before wound closure.
  Other Names: Isotonic saline
  Arms: 0.9% normal saline

SUMMARY:
The purpose of this study is to evaluate the efficacy of periarticular injection with 0.25% bupivacaine for controlling pain after total knee replacement to improve the quality of post-operative care.

DETAILED DESCRIPTION:
Compare post operative pain control after total knee replacement by periarticular injection with 0.25% bupivacaine compare with 0.9% normal saline.

ELIGIBILITY:
Inclusion Criteria:

* primary osteoarthritis patients undergoing total knee replacement at Siriraj Hospital
* BMI between 20-35
* having a full understanding of the question in this trial

Exclusion Criteria:

* allergy to NSAIDs, Acetaminophen, Bupivacaine
* blood creatinine more than 1.5 mg/dl or creatinine clearance less than 60 mL/min
* abnormal liver function
* previous surgery on the knee undergoing total knee replacement
* patient could not receive spinal anesthesia

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Post operative pain | 96 hour post operation
  Measure by Visual analog scale scores and morphine consumption

SECONDARY OUTCOMES:
Complication of Morphine consumption | 96 hour post operation
  nausea, pruritis, urinary retention and constipation

CONTACTS AND LOCATIONS:
Overall Officials: Keerati Chareancholvanich, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Mehrotra C, Remington PL, Naimi TS, Washington W, Miller R. Trends in total knee replacement surgeries and implications for public health, 1990-2000. Public Health Rep. 2005 May-Jun;120(3):278-82. doi: 10.1177/003335490512000310. PMID 16134568
- [Background] Akyol O, Karayurt O, Salmond S. Experiences of pain and satisfaction with pain management in patients undergoing total knee replacement. Orthop Nurs. 2009 Mar-Apr;28(2):79-85. doi: 10.1097/NOR.0b013e3181945f62. PMID 19339865
- [Background] Singelyn FJ, Deyaert M, Joris D, Pendeville E, Gouverneur JM. Effects of intravenous patient-controlled analgesia with morphine, continuous epidural analgesia, and continuous three-in-one block on postoperative pain and knee rehabilitation after unilateral total knee arthroplasty. Anesth Analg. 1998 Jul;87(1):88-92. doi: 10.1097/00000539-199807000-00019. PMID 9661552
- [Background] Toftdahl K, Nikolajsen L, Haraldsted V, Madsen F, Tonnesen EK, Soballe K. Comparison of peri- and intraarticular analgesia with femoral nerve block after total knee arthroplasty: a randomized clinical trial. Acta Orthop. 2007 Apr;78(2):172-9. doi: 10.1080/17453670710013645. PMID 17464603
- [Background] Vendittoli PA, Makinen P, Drolet P, Lavigne M, Fallaha M, Guertin MC, Varin F. A multimodal analgesia protocol for total knee arthroplasty. A randomized, controlled study. J Bone Joint Surg Am. 2006 Feb;88(2):282-9. doi: 10.2106/JBJS.E.00173. PMID 16452738
- [Background] Parvataneni HK, Shah VP, Howard H, Cole N, Ranawat AS, Ranawat CS. Controlling pain after total hip and knee arthroplasty using a multimodal protocol with local periarticular injections: a prospective randomized study. J Arthroplasty. 2007 Sep;22(6 Suppl 2):33-8. doi: 10.1016/j.arth.2007.03.034. Epub 2007 Jul 26. PMID 17823012
- [Background] Busch CA, Shore BJ, Bhandari R, Ganapathy S, MacDonald SJ, Bourne RB, Rorabeck CH, McCalden RW. Efficacy of periarticular multimodal drug injection in total knee arthroplasty. A randomized trial. J Bone Joint Surg Am. 2006 May;88(5):959-63. doi: 10.2106/JBJS.E.00344. PMID 16651569
- See also: Total knee replacement — http://www.nlm.nih.gov/medlineplus/kneereplacement.html
- See also: Bupivacaine information — http://www.rxlist.com/marcaine-drug.htm